CLINICAL TRIAL: NCT01742104
Title: Multicentric Observational Clinical Study on Quality of Life in Patients With Glaucoma in Italy
Brief Title: Multicentric Observational Study on Quality of Life in Glaucoma
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: IRFMN-OG1
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Primary Open-angle Glaucoma
Keywords: glaucoma; primary open-angle glaucoma; observational study; quality of life
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to evaluate the quality of life (QoL) of patients affected by Primary Open-Angle Glaucoma (POAG), using 2 QoL questionnaires:

1. Glaucoma Symptom Scale (GSS) and
2. National Eye Institute Visual Function Questionnaire (NEI-VFQ -25). The study will be conducted on patients with well known diagnosis of POAG (transversal phase) and on patients with first diagnosis of POAG (longitudinal phase).

DETAILED DESCRIPTION:
The study provides two levels of investigation, the first one (transversal phase), for all patients enrolled in the participating centers and the second one (longitudinal phase) conducted in a single cohort of patients with new diagnosis of POAG at enrollment.

The study will take part in around 20 centers specialized in glaucoma treatment and care, distributed throughout the Italian country area. The study aims to recruit a total of 3000 patients, around 200 of which with early diagnosis: they will represent the longitudinal cohort.

The frequency of visits and the type of examinations will follow the normal clinical practice.

The transversal phase consists of a single visit in which all socio-demographic and clinical characteristics of patients will be collected; during this visit patients will receive the NEI-VFQ 25 and the GSS questionnaires for measuring QoL (they have be filled in by the patient himself). For newly diagnosed patients, data collected during this visit will be consider as baseline, then they will enter in the longitudinal phase and will underwent two subsequent visits, the first one after about 6 months from baseline and the second one after a further 6 months (12 months from baseline). During the two subsequent visits the same data as the baseline will be collected, excluding for the socio-demographic data.

Patients will underwent examinations and therapy suitable for their disease treatment, based on physician judgment and according to the normal clinical practice.

All patient data will be collected on Case Report Form(CRF). All data contained in the CRF and in the QoL questionnaires, will be entered into an electronic database and will be checked in order to assess the plausibility, internal consistencies, errors or missing values. For each missing/loose/illegible/wrong data a request for clarification will be automatically generated by the system; it will be named "Query Form" and will be sent to the investigator for answers. At the end of the validation process, the database will be "frozen" and it will be used for statistical analysis.

The data were collected in an absolutely anonymous way. No data can be traced back up to the patient personal information or history.

All patients enrolled in the study, except for those with inclusion/exclusion criteria violations, will be considered in the statistical analysis.

The general characteristics of the study sample will be described. Qualitative variables will be described by means of the absolute and relative frequencies calculation, those quantitative with mean, standard deviation, quartiles, minimum, maximum, number of observations.

With regard to the QoL scale, the total score and subscale will be calculated. The same approach will be used within subgroups defined on the basis of socio-demographic and clinical characteristics.

As per the calculation of the sample size, it is estimated that at present in Italy there are 500,000 patients affected by glaucoma and about 50 centers specialized in the disease treatment.

A sample of 3000 patients with POAG and the involvement of at least 20 centers specialized in the glaucoma treatment are considered to be a representative estimation of reality in the Italian coutry area.

With a sample size of at least 3000 patients it is possible to calculate the 95%confidence interval of the estimated value of any parameter collected with an inaccuracy who not exceed 3.6%.

It is assumed that it will be possible to isolate about 200 patients in first diagnosis, in which the time course of the QOL scales scores will be described for the entire cohort and into predetermined patient subgroups.

For a successful implementation of the procedures required by the study the following activities are provided:

* Start-up and follow-up meetings, with the aim of sharing operating procedures, training the investigators to use the study tools for the collection of data and following-up study issues;
* Project dedicated Help Desk.

This study will be conducted according to AIFA March 20, 2008, "Guidelines for the classification and management of observational studies on drugs" and the principles expressed in the guidelines for the 'Good Epidemiology Practice' (GEP) in force in Europe.

A patient's informed consent and a consent to the processing of their data, signed by each patient, will be obtained before the study entry.

ELIGIBILITY:
Inclusion Criteria:

Patients with instrumental diagnosis of POAG, already being treated at the center or at the time of diagnosis

* Age > 18 years
* Ability to understand and answer to the questionnaires provided by the study
* Written consent to the processing of personal data.

Exclusion criteria:

* Female patients who are pregnant, breast-feeding or plan to become pregnant, or female patients of childbearing potential not using reliable means of birth control
* Concurrent abuse of alcohol and drugs
* Concurrent participation in any other clinical trial that tests drugs / medical devices within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary open-angle glaucoma (POAG).
Sampling Method: Non-Probability Sample
Enrollment: 3226 (Actual)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaires | up to 12 months
  National Eye Institute Visual Function Questionnaire (NEI-VFQ-25 - Italian Version, Jan 2003) Glaucoma Symptom Scale (GSS - Italian Version, April 2011)

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Quaranta, Professor MD, Principal Investigator — Università di Brescia - Italy
Locations (21):
- Italy (21):
  - Clinica Oculistica - Ospedale S. Salvatore, L’Aquila, AQ
  - U.O.Oftalmologia - Policlinico di Bari, Bari, BA
  - U.O. Oftalmologia Universitaria - Policlinico S. Orsola Malpighi, Bologna, BO
  - Dipartimento di Oftalmologia e Scienze Visive, Centro per lo studio del glaucoma - Spedali Civili, Brescia, BS
  - Reparto di Oculistica-Azienda Ospedaliera di Desenzano del Garda, Desenzano del Garda, BS
  - U.O. Oculistica - Ospedale Civile S. Giovanni di Dio, Cagliari, CA
  - Dipartimento Scienze per la Salute, Sezione Farmacologia Oculare - Università del Molise - Clinica Villa Maria,, Campobasso, CB
  - Clinica Oftalmologica-Ospedale Clinicizzato SS. Annunziata, Chieti, CH
  - U.O. Clinica Oculistica- A.O. Universitaria Policlinico Vittorio Emanuele, Catania, CT
  - U.O. Oculistica - Azienda Ospedaliera Universitaria Mater Domini, Catanzaro, CZ
  - Clinica Oculistica - Azienda Ospedaliera Ospedale San Martino, Genova, GE
  - U.O. Oculistica, Fondazione IRCCSS Ca' Granda Ospedale Maggiore Policlinico - Regina Elena, Milan, MI
  - Dipartimento Testa-Collo, Clinica Oculistica - Ospedale San Paolo, Milan, MI
  - Presidio Unico IRCCS S. Luca/S. Michele - Istituto Auxologico Italiano, Milan, MI
  - Clinica Oculistica - Azienda Ospedaliera Universitaria, Parma, PR
  - Clinica Oculistica - Fondazione IRCCS policlinico San Matteo, Pavia, PV
  - Struttura Complessa di Oculistica - Azienda Ospedaliera Arcispedale S. Maria Nuova, Reggio Emilia, RE
  - U.O.C. di Oculistica - Fondazione Policlinico Tor Vergata, Roma, RM
  - U.O. C. di Oftalmologia - Azienda Ospedaliera Universitaria S. Maria delle Scotte, Siena, SI
  - Clinica Oculistica dell'Università di Torino, Torino, TO
  - Clinica Oculistica - Azienda Ospedaliera Universitaria, Ospedali Riuniti, Trieste, TS

REFERENCES:
- [Derived] Riva I, Legramandi L, Katsanos A, Oddone F, Rulli E, Roberti G, Quaranta L; Italian Study Group on QoL in Glaucoma. Influence of Sociodemographic Factors on Disease Characteristics and Vision-related Quality of Life in Primary Open-angle Glaucoma Patients: The Italian Primary Open Angle Glaucoma Study (IPOAGS). J Glaucoma. 2018 Sep;27(9):776-784. doi: 10.1097/IJG.0000000000000989. PMID 29781833